CLINICAL TRIAL: NCT06844994
Title: Comparative Effects of Manual Diaphargmatic Technique Versus Lateral Coastal Breathing Exercise on Dyspnea, Chest Expansion and Functional Capacity Among COPD Patients.
Brief Title: Effects of Manual Diaphragmatic Technique Versus Lateral Coastal Breathing Exercises Among COPD Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0323 Maliha
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: COPD
Keywords: chronic obstructive pulmonary disease; Lung disease; Dysnea; Chronic airflow obstruction; Respiratory muscle training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Manual Diaphragmatic Technique
  Interventions: Other: Manual Diaphragmatic Technique
- Group B (Active Comparator): Lateral Coastal Breathing Exercises
  Interventions: Other: Lateral Coastal Breathing

INTERVENTIONS:
Other: Manual Diaphragmatic Technique — The intervention will be given 3 days per week for up to 6 weeks starting assessment with modified Borg scale questionnaire will be asked from the patient to evaluate the patient's dyspnea level. The patient at first will be asked to do 5-6 diaphragmatic breathing in upright position and then will be asked to breathe with the breather device after complete inhalation the patient will blow hard in the device. The patient will be asked to inhale and then hold for 2-3 second and breathe out through the device with the 3 sets with each set including 8 repetitions same cycle with relaxed diaphragmatic breathing between each set
  Arms: Group A
Other: Lateral Coastal Breathing — The group B will be the lateral coastal breathing that will be given 2 times a day, 3 days per week for up to 6 weeks. The patient will be asked by practitioner to perform 4 to 5 times lateral coastal breathing in suitable sitting or lying position
  Arms: Group B

SUMMARY:
Chronic obstructive pulmonary disease is a common, preventable as well treatable disorder, which is also one of the main reasons of high mortality and morbidity characterized by irreversible airflow limitation and has respiratory system involved. The aim of this study is to evaluate the comparative effects of manual diaphragmatic technique and lateral coastal breathing on COPD patients, that these exercises will have beneficial effects or not on COPD patients. Manual diaphragmatic technique and lateral coastal breathing will increase the functional capacity and relieve the symptoms dyspnea, enhance the chest wall expansion.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial to determine the effects of both techniques on COPD patients and disease severity in patients who falls into the inclusion criteria, who are willing to participate, patients with age limit between 45 to 65 years, GOLD stage II, and patients will be excluded who have cardiac disease, abdominal or thoracic surgeries and in critical condition by taking sample of patients through non probability convenient sampling and randomly allocating them to two groups A and B out of which A will receive manual diaphragmatic techniques, B will receive lateral coastal breathing exercise up to the duration of 2 times a day, 3 days per week for up to 3 weeks. Pre and post exercise outcomes will be assessed. The data will be analyzed through SPSS 26

ELIGIBILITY:
Inclusion Criteria:

Age 45-65 years(12). Both gender female and male. Patients willing to be the part of the research. Patients with moderate level of COPD Patients with GOLD II stage(13). Patients who response to bronchodilators Patients with history of smoking(14).

Exclusion criteria:

Patients having other cardiac diseases. Patients having thoracic or abdominal surgeries. Exacerbation of symptoms before or during study. Inability of Patient to understand instructions due to mental disorder Lack of medical record Coronary artery disease (coronary angiography with stenting or bypass) Malignant tumor Patients with gastrointestinal abnormalities Patients who are in critical condition

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female and male
Enrollment: 58 (Actual)
Dates: Start 2024-11-26 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
Measuring Tape | 6th week
  Measuring tape is used for chest wall measurement during inhalation and exhalation to compare differences
6 Mile Walk Test | 6 weeks
  6 mile walk test is used to perform to check functional capacity of the patient, it helps in assessment of the physical functional performance at baseline and post intervention, 6MWT will be performed inside the corridor on flat surface, the patients will be guided to walk on their own pace.
Modified Borg Scale | 6 Weeks
  Modified borg scale questionnaire will be asked from the patient to evaluate the patient's dyspnea level. Peak flow meter It is a handheld device that measures patient ability to push air out of your lungs, it is very useful in screening patients who have respiratory disorders and depicts the reliable respiratory state of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Qurat ul Ain, MS, Principal Investigator — Riphah International University
Locations (1):
- Ittefaq Hospital (Trust) Lahore., Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nair A, Alaparthi GK, Krishnan S, Rai S, Anand R, Acharya V, Acharya P. Comparison of Diaphragmatic Stretch Technique and Manual Diaphragm Release Technique on Diaphragmatic Excursion in Chronic Obstructive Pulmonary Disease: A Randomized Crossover Trial. Pulm Med. 2019 Jan 3;2019:6364376. doi: 10.1155/2019/6364376. eCollection 2019. PMID 30719351
- [Background] Similowski T, Yan S, Gauthier AP, Macklem PT, Bellemare F. Contractile properties of the human diaphragm during chronic hyperinflation. N Engl J Med. 1991 Sep 26;325(13):917-23. doi: 10.1056/NEJM199109263251304. PMID 1881417
- [Background] Siatras TA, Mittas VP, Mameletzi DN, Vamvakoudis EA. The duration of the inhibitory effects with static stretching on quadriceps peak torque production. J Strength Cond Res. 2008 Jan;22(1):40-6. doi: 10.1519/JSC.0b013e31815f970c. PMID 18296954
- [Background] Wada JT, Borges-Santos E, Porras DC, Paisani DM, Cukier A, Lunardi AC, Carvalho CR. Effects of aerobic training combined with respiratory muscle stretching on the functional exercise capacity and thoracoabdominal kinematics in patients with COPD: a randomized and controlled trial. Int J Chron Obstruct Pulmon Dis. 2016 Oct 28;11:2691-2700. doi: 10.2147/COPD.S114548. eCollection 2016. PMID 27822031
- [Background] Heneghan NR, Adab P, Balanos GM, Jordan RE. Manual therapy for chronic obstructive airways disease: a systematic review of current evidence. Man Ther. 2012 Dec;17(6):507-18. doi: 10.1016/j.math.2012.05.004. Epub 2012 Jun 15. PMID 22703901